CLINICAL TRIAL: NCT05451433
Title: The Effect of Saccharomyces Boulardii in Clinical Presentation and Quality of Life Patient With IBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Marcellus Simadibrata, Prof. PhD., SpPD, KGEH, Professor, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-03-0280
Record Dates: First submitted 2022-06-22; First posted 2022-07-11 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Get intervention drug Normagut capsule twice a day
  Interventions: Drug: Saccharomyces Boulardii 250 MG
- Control Group (Placebo Comparator): Get placebo capsule twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saccharomyces Boulardii 250 MG — Normagut capsule twice a day
  Other Names: Normagut
  Arms: Intervention Group
Drug: Placebo — Placebo capsule twice a day
  Arms: Control Group

SUMMARY:
This study aims to compare the effectiveness of Saccharomyces Boulardii vs Placebo in patient with Irritable Bowel Syndrome

DETAILED DESCRIPTION:
This study aims to compare the effectiveness of Saccharomyces Boulardii vs Placebo in patient with Irritable Bowel Syndrome within timeframe of study 28 days and then will be examined the outcome as the improvement quality of life

ELIGIBILITY:
Inclusion Criterias:

* 18 years or older
* diagnosed with IBS based on ROME IV criteria
* agree to be participant by signing inform consent

Exclusion Criteria:

* patient who does not want to sign the inform consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement quality of life within 29 days | 29 days
  Measuring quality of life using questionnaire IBS-QOL from 0-100, the higher the score, the better the outcome.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol